CLINICAL TRIAL: NCT03773159
Title: Development of a Device for Evaluating Primary Hemostasis Under Whole Blood Flow Conditions
Acronym: INDONESIA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: De MAISTRE ANR 2017
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Von Willebrand Diseases; Major Constitutional Thrombopathy; Patient on Antiplatelet Drugs
MeSH Terms: conditions — von Willebrand Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with von Willebrand disease or major constitutional thrombopathy or patients on antiplatelet drugs
  Interventions: Biological: Blood sampling
- Controls: Blood donors at the French blood establishment in Burgundy Franche-Comté
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — 4 citrated/PPACK tubes and 1 EDTA tube maximum

SUMMARY:
Currently, the exploration of primary hemostasis (a physiological phenomenon used to stop bleeding) is imperfect because it is based on targeted tests for platelets or von Willebrand factor, without taking into account blood flow and other blood cells (red and white blood cells). Tests for whole blood and flow conditions exist, but there is currently no test that comes close to actual physiological conditions.

An exploration of whole blood haemostasis in a device that is similar to a blood vessel and at different flow conditions (venous and arterial) could help to better identify the risk of bleeding in predisposed patients (von Willebrand factor deficiency, antiplatelet therapy).

The objective of the study is to evaluate the performance of this new hemostasis test in whole blood and under flow conditions.

Participation in the study is ad hoc and is limited to adding a maximum of 4 citrated tubes (20 mL or the equivalent of 4 teaspoons) and 1 EDTA tube (5mL) to a routine blood sample (for patients) or during blood donation (for controls).

ELIGIBILITY:
Inclusion Criteria:

* person who has given oral consent
* adult
* blood donor at EFS Bourgogne Franche-Comté
* or patient with von Willebrand disease or major constitutional thrombopathy followed by the Resource and Competence Centre (CRC) - Constitutional Hemorrhagic Diseases of Dijon or Besançon
* or patient on antiplatelet drugs consulting for thrombosis at the Dijon Bourgogne or Besançon Hospital

Exclusion Criteria:

* a person who is not affiliated to or not a beneficiary of national health insurance
* person subject to court-ordered protection (curatorship, guardianship)
* pregnant, parturient or breastfeeding woman
* a person who is unable to consent
* person on anti-inflammatory treatment and serotonin reuptake inhibitor antidepressants (platelet function disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with von Willebrand disease or major constitutional thrombopathy or patient on antiplatelet drugs
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Repeatability and reproducibility of the result in controls | Baseline
Detection of antiplatelet or von Willebrand factor deficiency/major constitutional thrombopathy | Baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - CHU Dijon Bourgogne, Dijon